CLINICAL TRIAL: NCT07250581
Title: Endoscopic Discectomy With Repair of Annulus Fibrosus Versus Discectomy Alone for Lumber Disc Herniation:A Prospective Multicenter Randomized Controlled Trial
Brief Title: A Randomized Trial of Annular Repair With Discectomy Versus Discectomy Alone for Lumbar Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); The Third Xiangya Hospital of Central South University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, maxuexiao, Endoscopic Discectomy with Repair of Annulus Fibrosus versus Discectomy Alone for Lumber Disc Herniation:A prospective Multicenter Randomized Controlled Trial, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QYFYEC2025-136
Record Dates: First submitted 2025-09-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Intervertebral Disc Herniation
Keywords: Annulus fibrosus repair; Lumbar intervertebral disc herniation; Spinal endoscopy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Annulus fibrosus repair (Experimental): Annulus fibrosus repair, Suture the incision of the annulus fibrosus
  Interventions: Procedure: Repair of the annulus fibrosus
- Non-annulus fibrosus repair (No Intervention): Non-annulus fibrosus repair, Do not suture the incision of the annulus fibrosus

INTERVENTIONS:
Procedure: Repair of the annulus fibrosus — Suture the incision of the annulus fibrosus
  Arms: Annulus fibrosus repair

SUMMARY:
The goal of this study is to explore the indications and application scope of spinal endoscopy combined with annulus fibrosus repair technology, with a focus on verifying the effectiveness of annulus fibrosus suture technology and evaluating its safety, so as to further support the promotion of annulus fibrosus repair technology in patients with lumbar disc herniation.

DETAILED DESCRIPTION:
1. Background Lumbar Disc Herniation (LDH) is a significant clinical and public health issue, particularly due to its high incidence and impact on working-age populations. It is a leading cause of non-fatal health loss globally. While conservative management is first-line, surgery is indicated for refractory cases. Among surgical options, endoscopic discectomy has emerged as a superior minimally invasive technique, offering advantages like minimal trauma, rapid recovery, and preserved spinal stability compared to open surgery or fusion.

   However, a key limitation of standard endoscopic discectomy is the residual defect in the annulus fibrosus (AF) after nucleus pulposus removal. This defect is a significant risk factor for postoperative recurrence, as residual disc material can re-herniate. Larger defects (≥6mm) are associated with significantly higher recurrence and reoperation rates. Annulus repair techniques, initially attempted in open surgery with limited success due to extensive tissue disruption, hold renewed promise in the minimally invasive endoscopic context. The recent development of dedicated endoscopic AF suture devices in China enables precise repair through the endoscope, potentially reducing recurrence and postoperative neural complications by restoring AF integrity, minimizing scar adhesion, and containing inflammatory mediators.

   Preliminary clinical application of this AF suture technique in over 12,000 cases suggests it adds only minimal time (~8 minutes) to the procedure while offering significant potential benefits. This study aims to rigorously evaluate the safety and efficacy of endoscopic discectomy combined with AF repair versus discectomy alone through a prospective, multicenter, randomized controlled trial (RCT).
2. Study Objectives and Significance Primary Objectives:To evaluate the efficacy of AF repair in reducing the postoperative recurrence rate of LDH.To assess the safety of AF repair by comparing perioperative complications and early postoperative pain exacerbation between the suture and control groups.

   Significance:This study will provide high-quality, multicenter RCT data to clarify the indications, technical nuances, clinical outcomes, and recurrence prevention effect of endoscopic AF suture. The findings will support the standardization and scientific application of this promising technology, offering valuable evidence for clinicians and patients in selecting optimal treatment strategies, particularly for young and active patients seeking rapid recovery and long-term durability.
3. Study Design and Methods Study Type: Prospective, multicenter, randomized controlled trial. Study Population:Participants: Patients aged 12-65 years diagnosed with symptomatic LDH from multiple participating centers.

Inclusion Criteria:

Age 12-65, any gender. Confirmed diagnosis of LDH. Non-calcified herniation type. Preoperative MRI shows Pfirrmann grade I-II disc degeneration. Failure of ≥6 months conservative treatment with significant impact on quality of life.

Willing and able to provide informed consent and comply with long-term follow-up.

Exclusion Criteria:

Concomitant lumbar spondylolisthesis, instability, or other significant spinal pathologies.

Previous lumbar spine surgery. Major systemic diseases contraindicating surgery. Conditions potentially affecting healing (e.g., malnutrition, bone metabolic diseases, autoimmune diseases).

Inability to adhere to follow-up schedule.

Intervention and Groups:Eligible patients will be randomly assigned to one of two groups:

Intervention Group: Endoscopic Discectomy + Annulus Fibrosus Repair. Control Group: Endoscopic Discectomy alone. Randomization: Randomization will be performed using PASS 11.0 generated random sequence after informed consent and baseline assessment, based on order of enrollment.

Outcome Measures:

Primary Outcomes:

Surgical success rate (successful completion of AF suture). Recurrence rate (re-herniation at the operated level) at short-term and long-term follow-up.

Postoperative efficacy: assessed by Visual Analog Scale (VAS) for back/leg pain, Japanese Orthopaedic Association (JOA) score, and Oswestry Disability Index (ODI).

Reoperation rate. Postoperative inflammatory markers (e.g., CRP, Procalcitonin).

Secondary Outcomes:

Incidence of nerve injury (sensory/motor). Incidence of bleeding/hematoma. Overall complication rate (e.g., infection, dural tear). Postoperative infection rate.

Data Collection and Follow-up:

Data collected includes demographic details, perioperative parameters (surgical level, time, blood loss, hospital stay), clinical scores (VAS, ODI, JOA), imaging data (herniation size, AF defect size, spinal canal area), and laboratory tests. Follow-up assessments are scheduled at 1, 3, 6, and 12 months postoperatively. Imaging follow-up includes MRI at 3 months, CT at 6 months, and both CT/MRI at 12 months.

Statistical Analysis:

Data will be managed using an Electronic Data Capture (EDC) system and analyzed with SPSS 25.0. Appropriate descriptive statistics will be used. Group comparisons for continuous variables will use t-tests or Mann-Whitney U tests, and chi-square tests for categorical variables. Repeated Measures ANOVA will analyze longitudinal data. Missing data will be handled with appropriate imputation methods and sensitivity analysis. A significance level of α=0.05 (two-sided) will be used.

Sample Size Calculation:

Based on an assumed recurrence rate of 5% in the control group and 2.4% in the intervention group, with α=0.05 and 90% power, a sample size of 224 is required. Accounting for a potential 20% dropout rate, the total target sample size is 300 patients. The lead center (Qingdao University Affiliated Hospital) will contribute approximately 100 patients.

Participating Centers (Multicenter):

The study involves one primary center and nine participating centers across China, each led by a principal investigator:

Primary Center: The Affiliated Hospital of Qingdao University. Participating Centers: Include Qilu Hospital of Shandong University, Shandong Provincial Hospital, Peking Union Medical College Hospital, The First Affiliated Hospital of Harbin Medical University, The First Affiliated Hospital of Wenzhou Medical University, The Third Xiangya Hospital of Central South University, The Second Affiliated Hospital of Xi'an Jiaotong University, The Fourth Affiliated Hospital of Zhejiang University School of Medicine, among others.

Ethics and Quality Control:

The protocol will be submitted for ethical approval at each center. Investigators will receive standardized training on the AF suture technique and data management procedures. Data integrity, accuracy, and confidentiality will be ensured through rigorous quality control measures, including training, data validation rules, double data entry checks, and secure handling of identifiable information.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12 years old to 65 years old, gender not limited;
2. Diagnosed with Lumbar disc herniation;
3. Preoperative intervertebral disc MRI Pfirrmann grade I - II;
4. Conservative treatment is ineffective, and the symptoms significantly affect life;
5. Be able to cooperate with long-term follow-up and sign the informed consent form.

Exclusion Criteria:

1. Accompanied by lumbar spondylolisthesis, lumbar instability and other lumbar diseases, etc.
2. Previous history of lumbar spine surgery;
3. Those who have other major physical diseases and are unable to tolerate surgery;
4. Diseases such as malnutrition, abnormal bone metabolism, and autoimmune diseases that may affect the postoperative development process;
5. Unable to accept regular follow-up visitors

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Within one year
  The proportion of lumbar intervertebral disc protrusion recurring at the surgical segment within a certain period after surgery, including short-term recurrence and long-term recurrence.
Postoperative therapeutic effect | Within one year
  The change of the quality of life of postoperative patients was evaluated by using the VAS(Visual Analog Score), Zero to ten points indicates the degree of pain from mild to severe
Postoperative therapeutic effect | Within one year
  The change of the quality of life of postoperative patients was evaluated by using the JOA score(Japanese Orthopaedic Association), In the JOA score, a range from 0 to 29 points is interpreted as indicating a progression from poor to good.
Postoperative therapeutic effect | Within one year
  The change of the quality of life of postoperative patients was evaluated by using the ODI (Oswestry Disability Index), 0% represents the least severe condition, while 100% indicates the most severe condition.

SECONDARY OUTCOMES:
Nerve injury | Within one year
  The proportion of postoperative nerve injury, including cases of sensory and motor nerve injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, China

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT07250581/SAP_000.pdf